CLINICAL TRIAL: NCT02261376
Title: Effects of Age, Gender & Race on the Pharmacokinetics (PK)of DS-1971a
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DS1971-A-E103
Record Dates: First submitted 2014-10-01; First posted 2014-10-10 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2015-01

CONDITIONS: Healthy
Keywords: pharmacokinetics
MeSH Terms: interventions — DS-1971a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Caucasian men, aged 18-55 years (Experimental)
  Interventions: Drug: DS-1971a
- Caucasian men, aged 65 years or older (Experimental)
  Interventions: Drug: DS-1971a
- Japanese men, aged 18-55 years (Experimental)
  Interventions: Drug: DS-1971a
- Caucasian women, aged 18-55 years (Experimental)
  Interventions: Drug: DS-1971a

INTERVENTIONS:
Drug: DS-1971a — DS-1971a is supplied as a powder or crystals and will be given as an oral suspension with Bitrex® (taste masking agent). Each subject will receive a single oral dose of 200 mg DS 1971a .

SUMMARY:
This is an open label, non-randomised, single-dose, parallel-group study in 48 healthy subjects enrolled in 4 cohorts - Caucasian men, aged 18-55 years, Caucasian men, aged 65 years or older, Japanese men, aged 18-55 years, Caucasian women, aged 18-55 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers:

  * Cohort 1: Caucasian men, aged 18-55 years
  * Cohort 2: Caucasian men, 65 years and older
  * Cohort 3: Japanese men, aged 18-55 years
  * Cohort 4: Caucasian women, aged 18-55 years For the purpose of determining eligibility, age is calculated at the day of dose administration
* Caucasian subjects (Cohorts 1-2 and 4) must have 4 Caucasian grandparents.
* Japanese subjects (Cohort 3 only) must have 4 ethnically Japanese grandparents, have a Japanese passport, and have lived outside Japan for no longer than 5 years.
* Female subjects (Cohort 4 only) must be of non-childbearing potential, as follows:
* they must be post-menopausal (the last menstrual period was at least 12 months ago, and a follicle-stimulating hormone (FSH) test at screening confirms post menopausal status); or
* they must be surgically sterile, that is undergone hysterectomy, bilateral oophorectomy, bilateral salpingectomy and/or bilateral tubal ligation.
* A BMI in the range 18-30 kg/m2, inclusive, and weighing between 50 and 100 kg at screening.
* Willing to comply with all study restrictions, including the use of contraception, concomitant medication, and dietary and lifestyle restrictions.
* Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
* Have given written consent to participate after reading the information and consent form, and after having the opportunity to discuss the trial with the investigator or his/her delegate.

  9. Have given written consent to have his/her data entered into The Over-volunteering Prevention System (TOPS).

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG findings, or laboratory values that could interfere with the objectives of the study or the safety of the subject.
* Presence of history of acute or chronic illness, including (but not limited to) liver or kidney disease, hypertension, seizures, or any known impairment of endocrine, or other specific body-organ dysfunction.
* Presence or history of severe adverse reaction to any medicine.
* Presence or history of malignant disease.
* Acute or chronic infectious disease, including human immunodeficiency virus (HIV), hepatitis B virus (HBV) or C virus (HCV) infection.
* Surgery (eg stomach bypass) or medical condition that might affect absorption of medicines.
* Significant illness within 4 weeks before the dose of study medication.
* Participation in another clinical trial of a new chemical entity or a prescription medicine within the previous 3 months, or unwilling to abstain from participating in other clinical trials during the study and for 3 months after receipt of study medication.
* Participation in another clinical study with DS-1971a.
* Blood pressure (BP) and heart rate in semi-supine position at the screening examination outside the ranges 90-140 mm Hg systolic, 40-90 mm Hg diastolic; heart rate 40-100 beats/min. Subjects with Stage 1 hypertension (systolic 140-160 mmHg; diastolic 90-100 mmHg) may be enrolled provided they do not have evidence of end-organ damage, diabetes or a 10 year cardiovascular risk >20%.
* Abnormal ECG waveform morphology at screening that would preclude accurate measurement of the QT interval duration.
* Corrected QT interval (Fridericia's formula) (QTcF) interval duration > 430 msec for men or > 450 msec for women, obtained as an average from the measurements on duplicate screening ECGs.
* Estimated glomerular filtration rate (eGFR) < 80 mL/min/1.73 m2 (younger subjects, Cohorts 1, 3 and 4) or < 70 mL/min/1.73 m2 (older subjects, Cohort 2) or an absolute creatinine value above the upper limit of the normal range. eGFR will be estimated using the modification of diet in renal disease [MDRD] equation).
* Use of any prescription medicine or over the counter (OTC) medications, or herbal remedies (such as St John's wort), known to be strong inhibitors or strong inducers of cytochrome (CYP) enzymes (also known as CYP450 enzymes) during the 30 days before the dose of trial medication; use of any other prescription or OTC medicine (except as permitted), including dietary supplements or herbal remedies, during the 7 days before the first dose of trial medication.
* Consumption of certain foods or beverages before the dose and throughout the study period.
* Loss of more than 400 mL blood during the 3 months before the trial, e.g., as a blood donor.
* Abuse of drugs or alcohol during the 2 years before the first dose of study medication, or intake of more than 21 units of alcohol weekly (for men) or 14 units of alcohol weekly (for women).
* Smoking more than 10 cigarettes or ½ ounce of tobacco daily and unwilling to stop smoking during the study.
* Likely possibility that the volunteer will not cooperate with the requirements of the protocol.
* Objection by General Practitioner (GP) to volunteer entering the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) Profile of DS-1971a | 4 days after dose administered
  PK: plasma concentrations of DS-1971a, and derived PK parameters: Cmax, tmax, tlast, t½, AUC0-inf, AUClast, %AUCextr, λz, Vz/F and CL/F.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 4 days after dose administered
  Number and severity of events will be measured and reported.
changes in laboratory profile as a measure of safety and tolerability | 4 days after dose administered
  clinically significant changes in blood and urine will be measured and reported (haemoglobin (Hb), red blood cells (RBC), mean corpuscular volume (MCV), mean corpuscular Hb (MCH), mean corpuscular Hb concentration (MCHC), haematocrit (HCT), white blood cells (WBC) and differential, platelets, urea, creatinine, uric acid, eGFR (only at screening), total bilirubin, total protein, albumin, globulin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transpeptidase (gamma GT), glucose, phosphate, cholesterol, triglycerides, potassium, sodium, calcium, chloride)
change in ECG profile | 4 days after dose administered
  clinically significant changes in ECG profile (such as QTc, PR interval, Ventricular rate, QRS) will be measured and reported

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/